CLINICAL TRIAL: NCT01908127
Title: The Effect of Filmed Modelling on the Anxious and Cooperative Behaviour of 4-6 Years Old Children During Dental Treatment
Brief Title: Efficacy of Film Modelling in Paediatric Dentistry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zahedan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, mehrsa paryab, assisstant professor, Zahedan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 1382
Record Dates: First submitted 2013-07-17; First posted 2013-07-25 (Estimated); Results first posted 2014-01-20 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2013-12

CONDITIONS: Cooperative Behaviour; Dental Anxiety
Keywords: film modelling; dental anxiety; cooperative behaviour; children

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tell- show- do procedure (Active Comparator): Group I (Tell- Show- Do Group): Tell-Show-Do, prophylaxis with paste and rubber cap and fluoride therapy was performed by the dentist for each participant in the operation room.
  In the second session,injection of loal anesthesia solution including a mandibular alveolar nerve block technique and the occlusal cavity preparation was performed.
  Interventions: Behavioral: tell- show- do; Drug: injection of local anesthesia solution; Procedure: occlusal cavity preparation
- film modelling (Experimental): Group II (Filmed modelling Group): the children were directed to a quiet and comfort room to watch a film presented by a dental assistant. The film showed that the same procedure consisted of Tell-Show-Do, prophylaxis with paste and rubber cap and fluoride therapy was performed on a 5-years-old child model with a time of 20 minutes. The child in the film was cooperative and was reinforced by a reward at the end of the procedure.
  In the second session, injection of loal anesthesia solution including a mandibular alveolar nerve block technique and the occlusal cavity preparation was performed.
  Interventions: Behavioral: film modelling; Drug: injection of local anesthesia solution; Procedure: occlusal cavity preparation

INTERVENTIONS:
Behavioral: tell- show- do — Children came in the operation room. Tell-Show-Do, prophylaxis with paste and rubber cap and fluoride therapy was performed by the dentist for each participant to increase their familiarity with dental procedures. The duration of the appointment was about 20 minutes and constant for all children.
  Arms: tell- show- do procedure
Behavioral: film modelling — the children were directed to a quiet and comfort room to watch a film presented by a dental assistant. The film showed that the same procedure consisted of Tell-Show-Do, prophylaxis with paste and rubber cap and fluoride therapy was performed on a 5-years-old child model with a time of 20 minutes. The child in the film was cooperative and was reinforced by a reward at the end of the procedure.
  Arms: film modelling
Drug: injection of local anesthesia solution — A topical anesthesia and injection of local anesthesia solution using mandibular alveolar nerve block technique was performed by the dentist
Procedure: occlusal cavity preparation — the occlusal cavity was prepared for pulpotomy and restoration of the teeth

SUMMARY:
The aim of this study is to evaluate the effect of Filmed modelling in comparison with commonly used Tell-Show-Do technique on the anxious and cooperative behaviour of 4-6 years old children during dental practice.

DETAILED DESCRIPTION:
This randomized clinical trial study was approved by ethics committee of Zahedan University of Medical Sciences and conducted in pediatric clinic of Zahedan dental school in 2010.

Among the patients referred to the clinic, forty six children aged 4-6 years (±2 months) were selected according to the inclusion criteria. They had caries lesion in one of the primary mandibular molars needed the pulpotomy and restoration treatment. It was confirmed that they have no previous experience of hospitalization and dental visit. The children with systemic diseases and developmental disorders were excluded from the study. The examination was completed and the necessary radiographies were prescribed.

Each child's parent was asked to complete the informed consent and a questionnaire gathering demographic characteristics of the child and family. Then, the child was enrolled in one of the study groups based on simple random sampling model as follow:

Group I (Tell- Show- Do Group): Children came in the operation room. Tell-Show-Do, prophylaxis with paste and rubber cap and fluoride therapy was performed by the dentist for each participant to increase their familiarity with dental procedures. The duration of the appointment was about 20 minutes and constant for all children. At the end of the first visit, the child was rewarded and the date of the second treatment visit was set for one week later.

In the second session, the child was entered the operating room alone. A video-camera located on the top of the dental unit light pole under a covering cloth was focused on the child's head and hands and started to record child's behavior.

The required injection including a mandibular alveolar nerve block technique was performed by the dentist. The heart beat rate of each child was recorded manually before and following the injection by the dentist. Then, the occlusal cavity was prepared for pulpotomy and restoration of the teeth. The treatment protocol was the same for all the participants.

In all children, parameters such as the attending dentist, his assistant, the working environment, time and duration (30 minutes for each child) of work, and the type of dialogues were all the same. Care was taken to make sure that the children were not tired, hungry, or did not have a common cold.

Group II (Filmed modelling Group): the children were directed to a quiet and comfort room to watch a film presented by a dental assistant. The film showed that the same procedure consisted of Tell-Show-Do, prophylaxis with paste and rubber cap and fluoride therapy was performed on a 5-years-old child model with a time of 20 minutes which was cooperative and reinforced by a reward at the end of the procedure. The produced film had been approved by 3 pediatric dentists.

The second treatment session was set for one week later. Dental procedures, measurement of the heart rate and recording of the behaviors were all performed as in Group I.

The recorded video tapes of all children were independently evaluated by 2 pediatric dentists who were blind to the grouping of the children. Children's anxiety reactions and cooperative behaviors were scored based on Venham Scale and Frankle Index, respectively .The viewers were asked to rate the child's responses in two stages: At the injection of local anesthesia and at the beginning of the tooth preparation.

Statistical analysis Mean of heart rate measurements and behavioral ratings were used for statistical analyses. Data analysis was performed applying t-test method in package of statistical software (SPSS- 15). All statistical references were made at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* children aged 4-6 years
* caries lesion in one of the primary mandibular molars needs to pulpotomy and restoration treatment.

Exclusion Criteria:

* children with systemic diseases and developmental disorders
* previous experience of hospitalization

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2010-09; Primary Completion 2011-02 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: mehrsa paryab, Dr, Principal Investigator — dental school, tehran university of medical sciences
Locations (1):
- Zahedan Dental School, Zahedan, Iran

RESULTS

PARTICIPANT FLOW:
Recruitment Details: September 2010- December 2010 paediatric clinic of dental school, Zahedan University of Medical Sciences
Pre-assignment Details: The parents of four the enrolled children declined the participation in the study
Period: Overall Study
Arm/Group | Tell- Show- do Procedure | Film Modelling
Started | 23 | 23
Completed | 22 | 23
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tell- Show- do Procedure | Film Modelling | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23 | 23 | 46
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.9 (1.17) | 5 (1.17) | 4.95 (1.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 13 | 9 | 22
Region of Enrollment [Number; unit: participants]
  Iran, Islamic Republic of | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Behaviors of Children
Description: A video-camera was focused started to record child's behavior. The recorded video tapes were independently evaluated by 2 paediatric dentists who were blind to the grouping of the children. Children's anxiety reactions and cooperative behaviours were scored based on venham scale and Frankle Index ,respectively. quantification was performed at the injection of local anaesthesia and at the beginning of the tooth preparation. An average of both two time points scoring was used.
  Table 1: Venham 6-point Index 0 = Relaxed: 1 = Uneasy: 2 = Tense: 3 = Reluctant: 4 = Interference: 5 = Out of contact
  Table 2: Frankle 4-point Index
  1:Definitely Negative ( uncooperative,Refusal of treatment ) , 2:Negative ( some evidence of negative attitude but not pronounced) , 3:Positive ( Acceptance of treatment, at times cautious) , 4:Definitely Positive( Good rapport with the dentist)
Time Frame: participants followed for the duration of examination and treatment appointment, an expected average of 3 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tell- Show- do Procedure | Film Modelling
Number analyzed (Participants) | 22 | 23
units on a scale
  anxious behaviour quantification | 0.97 (0.73) | 1.09 (0.99)
  cooperative behaviour quantification | 2.95 (0.64) | 2.98 (0.67)

2. Secondary Outcome: Index of Heart Rate
Description: The heart rate of children was measured before the injection of local anesthesia solution to save a baseline data and it was also measured after the injection to assess the effect of this dental stress.
Time Frame: before and after the injection of local anesthesia solution
Measure: Mean (Standard Deviation); unit: beat per Min
Arm/Group | Tell- Show- do Procedure | Film Modelling
Number analyzed (Participants) | 22 | 23
beat per Min
  baseline heart rate | 99.27 (9.17) | 102.73 (12.37)
  heart rate after the injection | 110.40 (10.86) | 113 (13.86)

ADVERSE EVENTS:
Arm/Group | Tell- Show- do Procedure | Film Modelling
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 0/22 | 0/23

LIMITATIONS AND CAVEATS:
providing a quiet environment and patient sampling were the most important limitations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No